CLINICAL TRIAL: NCT07374432
Title: Full Speed Ahead: For Joyful Movement and Health
Acronym: fullspeed
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ann-Christin Eliasson, Professor, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2024-05809-01; Privat donations 3 500 000 SEK (Other: Karolinska Institutet)
Record Dates: First submitted 2025-11-18; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; Frame running; early intervention; children; mobility; physical activity
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Intervention Model Description: Singel subject design with 3 baseline before intervention and 3 follow up after intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): Frame running and gross motor training
  Interventions: Behavioral: Full speed ahead

INTERVENTIONS:
Behavioral: Full speed ahead — 12 weeks of daily training at home and 1 group training session /week including both Frame running and grossmotor training

SUMMARY:
The aim of this project is to implement and evaluate the effects of a mobility-focused training program, including the use of running frames, on gross motor function and physical activity levels in children aged 2-5 years with cerebral palsy. The hypothesis is that these children can improve their mobility with or without assistive devices, that the training program will influence their overall activity level, and that it will provide cardiovascular exercise leading to improved fitness and muscle development.

In previous studies, the investigators have observed positive health-related outcomes in older children. Recently, three-wheeled Frame Running bikes designed for very young children have become available; however, no research has been conducted on these devices or their potential effects in toddlers.

In this project, group training sessions will be offered to children aged 2-5 years. Participants will receive mobility and gait training with or without assistive devices, depending on individual needs. The three-wheeled Frame Running bike will be included as one training component, although participants may use other assistive aids as needed. Training is planned as play-based activities together with peers, for one hour per week over a 12-week period, complemented by home-based exercises.

ELIGIBILITY:
Inclusion Criteria:

GMFCS II-V

Exclusion Criteria:

severe intelectual disability

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-12-07 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function MEasure (GMFM) | From enrollment to the end of treatment at 3 month
  Measure gross motor function in children with CP from 6 month to 18 years, the scale ranging from 0-100 units, higher is better

SECONDARY OUTCOMES:
Sens motion, Accelerometry | From enrollment to the end of intervention at 3 months
  Measure physical activity in daily life

OTHER OUTCOMES:
Functional mobility scale (FMS) | From enrollment to the end of treatment at 3 months
  Measure childrens ability to walk on a 5 graded scale
Pediatric Evaluation of the Disability Inventory (PEDI- CAT) | From enrollment to the end of treatment at 3 month
  Mobility module measure childrens ability to move in the environment on a 0-100 scale
Time up and Go (TUG) | From enrollment to the end of treatment at 3 months
  Measure balans in standing and motion, mesaure in seconds
Goal Attainment scale (GAS) | From enrollment to the end of treatment at 3 month
  Measure individualized goals, based a a 5-graded scale
Ultra sound | From enrollment to the end of treatment at 3 months
  Measure the muscles thickness and form
Pediatrice Rehabilitation Intervention Measure of Engagement for Parents (Prime P) | From enrollment to the end of treatment at 3 month
  Descrieb the parents engagement in treatment
Service Provider-Rated Measure of Client Engagement (Prime SP) | From enrollment to the end of treatment at 3 month
  Describe the therapist's assessment of the child's engagement
Wrist-worn heart rate monitor | From enrollment to the end of treatment at 3 weeks
  Measure the pulse continously during certain period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Woman's and Children's health, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Patient data and we need to know more about the result